CLINICAL TRIAL: NCT05016778
Title: A Single Arm, Open Label Clinical Study of CAR-T Cells Targeting GPRC5D in the Treatment of Relapsed / Refractory Multiple Myeloma(POLARIS)
Brief Title: A Study of CAR-T Cells Targeting GPRC5D in the Treatment of r/r Multiple Myeloma
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Zhejiang University (Other)
Collaborators: OriCell Therapeutics Co., Ltd. (Industry)
Responsible Party: Principal Investigator, He Huang, Chief Physician, Zhejiang University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: POLARIS
Record Dates: First submitted 2021-06-06; First posted 2021-08-23 (Actual); Last update posted 2022-11-01 (Actual); Status verified 2022-10

CONDITIONS: Multiple Myeloma
Keywords: CAR-T; GPRC5D; Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment Group (Experimental): This is a open label, single arm clinical trial.
  Interventions: Drug: GPRC5D-CAR-T

INTERVENTIONS:
Drug: GPRC5D-CAR-T — After enrollment, subjects complete the PBMC apheresis, then complete the Lymphocyte clearance, and then receive the dose climbing test: 1×10e6/kg，3×10e6/kg，6×10e6/kg.

SUMMARY:
This is a single-arm, open-label, dose-escalation study to evaluate the safety, tolerability, cellular kinetics and initial efficacy of CAR-T cell therapy targeting GPRC5D in multiple myeloma subjects who have failed the standard treatments.

ELIGIBILITY:
Inclusion Criteria:

1. The subject can understand and have the ability to sign an informed consent form;
2. Male or female subjects, aged 18-75 years;
3. The expected survival period is not less than 12 weeks;
4. ECOG score ≤ 2 ;
5. Diagnosed as multiple myeloma according to the IMWG standard in 2018;
6. The expression of GPRC5D in bone marrow plasma cells is more than 20%, or it is positive in tumor tissue by immunohistochemistry. One of the following criteria must be detected:

   1. If IgG type MM, serum M protein ≥10g/L; if IgA, IgD, IgE or IgM type MM, serum M protein ≥5g/L;
   2. Or urine M protein level ≥200mg/24h;
   3. Or light chain type MM, serum free light chain (sFLC) ≥ 100mg / L and K/ λ FLC ratio is abnormal;
   4. Or there are extramedullary lesions;
7. Subjects who have received at least 3 different mechanism drugs (including chemotherapy, protease inhibitors, immunosuppressive agents, etc.) have failed treatments, or have progressed or recurred during the last treatment or within 6 months after the end of treatment ;
8. Lung function is normal, and oxygen saturation is greater than 92%;
9. No heart disease or coronary heart disease, echocardiogram showed normal diastolic function, left ventricular ejection fraction (LVEF) ≥50%, and no serious arrhythmia;
10. Liver function: TBIL<3×ULN, AST<2.5×ULN, ALT<2.5ULN;
11. Renal function: creatinine clearance rate (estimated by Cockcroft Gault formula) ≥ 30 mL/min;
12. The blood routine meets the following standards:

    1. Lymphocyte count>0.5×10e9/L;
    2. Neutrophils ≥1.0×10e9/L;
    3. Hemoglobin ≥80g/L;
    4. Platelet ≥75×10e9/L
13. From the use of study drug to 2 years after treatment, male subjects or female subjects of childbearing age must agree and be able to take effective contraceptive measures.

Exclusion Criteria:

1. Pregnant or breastfeeding;
2. HBsAg or HBcAb are positive, and the quantitative detection of HBV DNA in peripheral blood is more than 100 copies / L; HCV antibody and HCV RNA in peripheral blood are positive; HIV antibody positive; Syphilis antibody is positive in the first screening;
3. Any unstable systemic disease: including but not limited to unstable angina, cerebrovascular accident or transient cerebral ischemia (within 6 months before screening), myocardial infarction (within 6 months before screening), congestive heart failure (New York Heart Association [NYHA] classification ≥ grade III), severe arrhythmia with poor drug control, liver, kidney or metabolic diseases;
4. Had hypersensitivity or intolerance to any drug used in this study;
5. Patients who received anti-cancer chemotherapy or other medications within 2 weeks before screening;
6. Uncontrolled malignant tumors except MM, excluding malignant tumors that received radical treatment and no active disease was found within 3 years before enrollment;
7. Clinically significant central nervous system diseases, such as epilepsy, cerebrovascular ischemia/hemorrhage, dementia, cerebellar disease, psychosis, active central nervous system involvement or cancerous meningitis;
8. In the past two years, autoimmune diseases (such as Crohn's disease, rheumatoid arthritis, systemic lupus erythematosus) caused damage to terminal organs, or required systemic application of immunosuppressive or other drugs;
9. Severe active viral, bacterial or uncontrolled systemic fungal infections; Hereditary bleeding / coagulation diseases, history of non traumatic bleeding or thromboembolism, other diseases that may increase the risk of bleeding, etc;
10. Patients who received autologous hematopoietic stem cell transplantation (ASCT) within 8 weeks before screening, or who plan to undergo ASCT during the study period;
11. Patients received allogeneic stem cell therapy;
12. Any unsuitable to participate in this trial judged by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2021-06-08 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Dose limited toxicity (DLT) | From date of initial treatment to Day 28 post GPRC5D CAR-T infusion.
  Dose limited toxicity
AE and SAE | From admission to the end of the follow-up, up to 2 years
  Adverse event and serious adverse event

SECONDARY OUTCOMES:
Concentration of CAR-T cells | From admission to the end of the follow-up, up to 2 years
  In peripheral blood and bone marrow
Objective Response Rate, ORR | In 3 months of GPRC5D CAR-T cell infusion
  Proportion of subjects with complete or partial remission
Disease control rate, DCR | From Day 28 GPRC5D CAR-T infusion up to 2 years
  The percentage of patients with remission and stable disease after treatment in the total evaluable cases.
Duration of remission, DOR | 24 months post GPRC5D CAR-T cells infusion
  The time from the first assessment of remission or partial remission of the tumor to the first assessment of disease progression or death from any cause;
Progression-free survival, PFS | 24 months post GPRC5D CAR-Tcells infusion
  The time from cell reinfusion to the first assessment of tumor progression or death from any cause
Overall survival, OS | From GPRC5D CAR-T infusion to death，up to 2 years
  The time from the cell reinfusion to death due to any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Huang He, Principal Investigator — Hematology
Locations (1):
- The first affiliated hospital of medical college of zhejiang university, Hangzhou, Zhejiang, China

REFERENCES:
- [Derived] Zhang M, Wei G, Zhou L, Zhou J, Chen S, Zhang W, Wang D, Luo X, Cui J, Huang S, Fu S, Zhou X, Tang Y, Ding X, Kuang J, He XP, Hu Y, Huang H. GPRC5D CAR T cells (OriCAR-017) in patients with relapsed or refractory multiple myeloma (POLARIS): a first-in-human, single-centre, single-arm, phase 1 trial. Lancet Haematol. 2023 Feb;10(2):e107-e116. doi: 10.1016/S2352-3026(22)00372-6. PMID 36725117